CLINICAL TRIAL: NCT06933732
Title: The Effect of Virtual Reality Applications on Patient Outcomes and Satisfaction Before and After Total Knee Replacement: A Randomised Controlled Study
Brief Title: Effect of Virtual Reality on Patient Outcomes and Satisfaction in Total Knee Replacement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aykut Turgut (Other)
Responsible Party: Sponsor-Investigator, Aykut Turgut, Research Assistant, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-AT-02
Record Dates: First submitted 2025-03-02; First posted 2025-04-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Knee Replacement; Knee Replacement Surgery; Postoperative Pain, Acute; Anxiety, Preoperative; Pain Management; Virtual Reality
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Participants in this group will receive standard care, which includes preoperative education about the surgical process via an educational video and the completion of informed consent. No virtual reality intervention will be provided during their recovery.
- 2-Hour Postoperative VR Intervention (Experimental): Participants in this group will first watch an educational VR video about the surgery before the procedure. Two hours post-surgery, they will be exposed to a VR intervention featuring calming nature videos.
  Interventions: Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (2 hours)
- 4-Hour Postoperative VR Intervention (Experimental): Participants in this group will first watch an educational VR video about the surgery before the procedure. Four hours post-surgery, they will be exposed to a VR intervention featuring calming nature videos.
  Interventions: Device: Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (4 hours)
- 6-Hour Postoperative VR Intervention (Experimental): Participants in this group will first watch an educational VR video about the surgery before the procedure. Six hours post-surgery, they will be exposed to a VR intervention featuring calming nature videos.
  Interventions: Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (6 hours)

INTERVENTIONS:
Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (2 hours) — The Virtual Reality intervention involves participants wearing a VR headset at least one hour prior to their surgery to watch immersive, pre-recorded educational videos showing the operating room with a nurse explaining the process aimed at reducing pre-operative anxiety and nature videos with distraction effect after surgery for pain management. The intervention for pain management will be delivered 2 hours after surgery. The videos to be shown to patients will be limited to a maximum of 30 minutes. In addition, all participants will be reminded that they can remove the glasses or leave the study at any time.
  Arms: 2-Hour Postoperative VR Intervention
Device: Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (4 hours) — The Virtual Reality intervention involves participants wearing a VR headset at least one hour prior to their surgery to watch immersive, pre-recorded educational videos showing the operating room with a nurse explaining the process aimed at reducing pre-operative anxiety and nature videos with distraction effect after surgery for pain management. The intervention for pain management will be delivered 4 hours after surgery. The videos to be shown to patients will be limited to a maximum of 30 minutes. In addition, all participants will be reminded that they can remove the glasses or leave the study at any time.
  Arms: 4-Hour Postoperative VR Intervention
Device: Virtual Reality Intervention for Preoperative Anxiety and Postoperative Pain Management (6 hours) — The Virtual Reality intervention involves participants wearing a VR headset at least one hour prior to their surgery to watch immersive, pre-recorded educational videos showing the operating room with a nurse explaining the process aimed at reducing pre-operative anxiety and nature videos with distraction effect after surgery for pain management. The intervention for pain management will be delivered 6 hours after surgery. The videos to be shown to patients will be limited to a maximum of 30 minutes. In addition, all participants will be reminded that they can remove the glasses or leave the study at any time.
  Arms: 6-Hour Postoperative VR Intervention

SUMMARY:
This study aims to evaluate the effectiveness of virtual reality (VR) in managing preoperative anxiety and postoperative pain in patients undergoing total knee replacement. Investigators will assess the impact of preoperative VR training on anxiety levels, explore the effectiveness of relaxing and distracting VR videos for pain management after surgery, and determine the optimal timing for VR application by comparing different VR intervention times. Our goal is to identify how VR can improve both the emotional and physical recovery process for patients undergoing knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ASA score of 1, 2, or 3
* Elective unilateral total knee replacement surgery was planned,
* Patients who are able to read and write in Turkish

Exclusion Criteria:

* Using >30 mg of oral oxycodone or equivalent daily
* Long-term opioid use (>12 weeks)
* Substance use disorder
* Scheduled for emergency surgery
* Scheduled for revision surgery
* Requiring postoperative intensive care
* Patients with visual or hearing impairments
* Individuals experiencing motion-related nausea or dizziness
* History of stroke or dementia
* Pregnant or breastfeeding women
* Patients with a history of epilepsy or seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain Intensity as Measured by Visual Analogue Scale (VAS) at 2, 4, and 6 Hours After Surgery in Patients Receiving Virtual Reality Interventions. | Baseline (before VR intervention) and assessments at 2, 4, and 6 hours after surgery, with a 15-Minute wait after VR video completion before each pain assessment
  0 = No pain 10 = Worst pain possible

SECONDARY OUTCOMES:
Preoperative Anxiety Measured Using the State-Trait Anxiety Inventory-State (STAI-S) Scale | Baseline (just before the educational video) and post-video (immediately after the educational video, Day 1)
  Preoperative anxiety will be measured using the State-Trait Anxiety Inventory-State (STAI-S) scale, which is a validated tool for assessing temporary feelings of anxiety. Patients will complete the scale before undergoing any intervention or VR exposure. This measurement will provide an understanding of the patient's baseline anxiety level before the application of VR. This measurement will be taken twice: once before the patients view the educational videos and once after viewing them.
  Total scores range from 20 to 80. Higher scores = Higher levels of anxiety.
Change from Baseline in Virtual Reality Sickness as Measured by the Virtual Reality Sickness Questionnaire (VRSQ) | Baseline (just before the educational video) and post-video (immediately after the educational video, Day 1)
  The Virtual Reality Sickness Questionnaire (VRSQ) assesses the level of discomfort or sickness experienced by participants during or immediately after wearing the Virtual Reality headset.
  Total scores range from 0 to 15, with higher scores indicating higher levels of discomfort or sickness.
Patient Satisfaction as Measured by a 0-10 Numeric Rating Scale Post-Intervention | Postoperative, Day 1
  Patient satisfaction will be measured using a 0-10 Numeric Rating Scale (NRS), where 0 represents no satisfaction and 10 represents the highest level of satisfaction.
Change in Body Temperature (Celsius) from Baseline | Baseline (just before VR intervention) and 2, 4, or 6 hours post-surgery, depending on the assigned group.
Change in Heart Rate/min from Baseline | Baseline (just before VR intervention) and 2, 4, or 6 hours post-surgery, depending on the assigned group.
Change in Blood Pressure from Baseline (Systolic/Diastolic mmHg) | Baseline (just before VR intervention) and 2, 4, or 6 hours post-surgery, depending on the assigned group.
Change in Respiratory Rate/min from Baseline | Baseline (just before VR intervention) and 2, 4, or 6 hours post-surgery, depending on the assigned group.
Change in Blood Oxygen Saturation(%) from Baseline | Baseline (just before VR intervention) and 2, 4, or 6 hours post-surgery, depending on the assigned group.

OTHER OUTCOMES:
Postoperative Infection Incidence in Participants | Perioperative/Periprocedural
  The incidence of postoperative infections in participants from surgery until discharge. Infections will be identified based on clinical evaluation and standard medical criteria, and recorded for each participant.
Change in Hospital Stay Duration | Perioperative/Periprocedural
  The total duration of the hospital stay, including both preoperative and postoperative periods.
Change in Opioid Usage Postoperatively | Perioperative/Periprocedural
  The total amount of opioids used postoperatively, measured in standardized doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Aibu Izzet Baysal Training and Research Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be shared at this time, as it is considered important to first publish the data in the form of a manuscript.